CLINICAL TRIAL: NCT02989584
Title: A Pilot Safety Study and Single Arm Phase II Study of Gemcitabine and Cisplatin With Atezolizumab (MPDL3280A) in Patients With Metastatic and Muscle Invasive Bladder Cancer, Respectively
Brief Title: A Phase II Study of Atezolizumab in Combination With Cisplatin + Gemcitabine Before Surgery to Remove the Bladder Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-1428
Record Dates: First submitted 2016-12-02; First posted 2016-12-12 (Estimated); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Bladder Cancer; Metastatic Bladder Cancer; Urothelial Carcinoma
Keywords: bladder cancer; metastatic bladder cancer; atezolizumab; urothelial carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — atezolizumab; Gemcitabine; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- Atezolizumab, Gemcitabine, Cisplatin (Experimental): This is a two phase study with a single study arm for each phase.
  For Phase 1: Following enrollment participants will be treated with combination therapy on a 21 day cycle x 6 cycles. Gemcitabine (1000 mg/m2 on Day 1 and Day 8), cisplatin (70 mg/m2 on Day 1), and atezolizumab (1200 mg on Day 8) will be administered intravenously.
  Phase 2: Following enrollment participants will be treated with a single dose of atezolizumab alone followed by combination therapy on a 21-day cycle x 4 cycles, followed by a single dose of atezolizumab alone. Gemcitabine 1000mg/m2, cisplatin (70 mg/m2 on Day 1), and atezolizumab (1200 mg on Day 8) will be administered intravenously.
  Interventions: Drug: Atezolizumab; Drug: Gemcitabine; Drug: Cisplatin

INTERVENTIONS:
Drug: Atezolizumab
Drug: Gemcitabine
Drug: Cisplatin

SUMMARY:
The purpose of this study is to test the safety of the study drug, atezolizumab, when combined with the standard chemotherapy drugs, gemcitabine and cisplatin (or GC). This study will help researchers begin to understand whether combining GC with atezolizumab is better, the same, or worse than the usual approach of using GC alone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* ECOG Performance Status of 0 or 1
* Required Initial Laboratory Values within 14 days of enrollment:

  * Absolute Neutrophil Count ≥ 1500 cells/mm^3
  * Lymphocyte count ≥ 300/mm^3
  * Platelets ≥ 100,000 cells/mm^3
  * Hemoglobin ≥ 9.0 g/dL
  * Bilirubin ≤ 1.5 the upper limit of normal (ULN) for the institution For patients with known Gilbert's disease: bilirubin ≤ 3 x ULN
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 x ULN for the institution.

    * For patients in the metastatic cohort with documented liver or bone metastases: AST and/or ALT ≤ 5.0 x ULN
  * Alkaline phosphatase ≤ 2.5 x ULN for the institution

    * For patients in the metastatic cohort with documented liver or bone metastases: alkaline phosphatase ≤ 5 x ULN
  * If female of childbearing potential, urine pregnancy test is negative.
  * INR and aPTT ≤ 1.5 x ULN if not on therapeutic anticoagulation. Patients receiving therapeutic anticoagulation should be on a stable dose.

Phase I Cohort

* Archival tumor specimens must be submitted prior to enrollment. Samples collected from fine-needle aspiration, brushing, cell pellet from pleural effusion, bone metastases, and lavage are not acceptable. Acceptable samples include core-needle biopsies for deep tumor tissue (minimum of three cores) or excisional, incisional, punch, or forceps biopsies for cutaneous, subcutaneous, or mucosal lesions. If archival tissue is being used, representative urothelial carcinoma FFPE tumor specimens (tumor blocks or 30 unstained slides) must be provided. Patients with < 30 slides may be enrolled after discussion with the principal investigator. Primary or metastatic specimens may be submitted.
* Subject must agree to undergo two research-directed biopsies during treatment.
* The patient must have measurable disease according to RECIST v1.1 and must have one site amenable to biopsy that, in the opinion of the investigator and/or interventional radiologist, is likely to yield acceptable tumor sample for a core biopsy per the above pathology criteria.
* Life expectancy ≥ 12 weeks
* Histologically or cytologically confirmed urothelial carcinoma (confirmed at the enrolling institution) of the bladder, ureter, urethra, or renal pelvis. Patients with mixed histologies are required to have a predominant urothelial component as reviewed by the pathologist at the treating institution.
* Locally advanced (T4b, any N; any T, N2-3) or metastatic (M1) disease as determined by the treating investigator
* Estimated glomerular filtration rate ≥ 60 ml/min/1.73m2 using the CKD- EPI equation: eGFR = 141 x min(Scr/k, 1)a x max(Scr/k, 1)-1.209 x 0.993Age°x 1.018 [if female] x 1.159 [if black] Scr is serum creatinine, k is 0.7 for females and 0.9 for males, a is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/k or 1, and max indicates the maximum of Scr/k or 1

Phase 2 Cohort

* Pathology: Representative urothelial carcinoma FFPE tumor specimens (tumor blocks or 30 unstained slides). Patients with < 30 slides may be enrolled after discussion with the principal investigator.
* Muscle invasive urothelial carcinoma of the bladder histologically confirmed at the enrolling institution. (Urothelial carcinoma invading into the prostatic stroma with no histologic muscle invasion is allowed provided the extent of disease is confirmed via imaging and/or EUA.)
* Clinical stage T2-4a;N0/X;M0
* Medically appropriate candidate for radical cystectomy, as per MSK or participating site Attending Urologic Oncologist
* Estimated glomerular filtration rate ≥ 60 ml/min/1.73m2 using the CKD- EPI equation: eGFR = 141 x min(Scr/k, 1)a x max(Scr/k, 1)-1.209 x 0.993Age°x 1.018 [if female] x 1.159 [if black] Scr is serum creatinine, k is 0.7 for females and 0.9 for males, a is -0.329 for females and -0.411 for males, min indicates the minimum of Scr/k or 1, and max indicates the maximum of Scr/k or 1

Exclusion Criteria:

* Evidence of NYHA functional class III or IV heart disease
* Serious intercurrent medical or psychiatric illness, including serious active infection
* Preexisting sensory grade ≥ 2 neuropathy
* Preexisting grade ≥ 2 hearing loss
* Major surgical procedure within 28 days prior to Cycle 1, Day 1 or anticipation of need for a major surgical procedure during the course of the study. Transurethral resection or other urinary tract diagnostic procedures, excisional biopsy, or MediPort placement, are NOT defined as major surgical procedures.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack
* Ongoing cardiac dysrhythmias of NCI CTCAE Version 4.0 grade ≥ 2. However, stable atrial fibrillation controlled medically or with a device (e.g. pacemaker) or prior ablation is allowed.
* History of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness
* Concurrent treatment on another clinical trial; supportive care trials or non-treatment trials, e.g. QOL, are allowed
* Pregnancy, lactation, or breast-feeding. Patients must be surgically sterile, postmenopausal, or must agree to use effective contraception during the period of therapy and for 5 months after the last dose of atezolizumab. The definition of effective contraception will be based on the judgment of the principal investigator or a designated associate. Male patients must be surgically sterile or agree to use effective contraception. Male patients will be encouraged to notify the study team if their female partner becomes pregnant while on study.
* History of autoimmune disease, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, Wegener's granulomatosis, vascular thrombosis associated with antiphospholipid syndrome, Sjogren's syndrome, Guillain-Barre syndrome, multiple sclerosis, systemic vasculitis, or glomerulonephritis.

  * Patients with history of autoimmune related hypothyroidism on stable dose of thyroid replacement hormone may be eligible for this study
  * Patients with controlled Type I diabetes mellitus on a stable dose of insulin may be eligible for this study
* History of idiopathic pulmonary fibrosis, pneumonitis (including drug induced), organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia, etc.), or evidence of active pneumonitis on screening chest computed tomography (CT) scan

  * History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Patients with active hepatitis B virus (HBV, chronic or acute, defined as having a positive hepatitis B surface antigen [HBsAg] test at screening) or hepatitis C antibody

  * Patients with past HBV infection or resolved HBV infection (defined as the presence of hepatitis B core antibody [HBc Ab] and absence of HBsAg) are eligible. HBV DNA must be obtained in these patients prior to Cycle 1, Day

    1 and confirmed to be negative.
  * Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Active tuberculosis or BCG infection
* Severe infections within 4 weeks prior to Cycle 1, Day 1, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumonia
* Signs or symptoms of infection within 2 weeks prior to Cycle 1, Day 1. Abnormal urinalysis does not constitute signs/symptoms of infection unless urine culture obtained at screening grows ≥ 100,000 colonies of bacteria. Patients with an ileal conduit and a urinalysis and/or culture that are abnormal are eligible unless they have peripheral blood WBC > ULN, fever, or other symptoms suggestive of a urinary tract infection.
* Therapeutic oral or IV antibiotics within 2 weeks prior to Cycle 1, Day 1

  * Patients receiving prophylactic antibiotics (e.g., for prevention of a urinary tract infection or to prevent chronic obstructive pulmonary disease exacerbation) are eligible.
* Prior allogeneic stem cell or solid organ transplant
* Administration of intravesical bacillus Calmette-Guerin (BCG) within 4 weeks before Cycle 1, Day 1
* Administration of a live, attenuated vaccine within 4 weeks before Cycle 1, Day 1 or anticipation that such a live attenuated vaccine will be required during the study.

  * Influenza vaccination should be given during influenza season only (approximately October to March). Patients must not receive live, attenuated influenza vaccine (e.g., FluMist ®) within 4 weeks prior to Cycle 1, Day 1 or at any time during the study.
* AEs from prior anticancer therapy that have not resolved to Grade ≤ 1 except for alopecia
* Bisphosphonate therapy for symptomatic hypercalcemia

  * Use of bisphosphonate therapy for other reasons (e.g., bone metastasis or osteoporosis) is allowed.
* Known clinically significant liver disease, including active viral, alcoholic, or other hepatitis; cirrhosis; and inherited liver disease
* Patients with a history of or active bone marrow disorders expected to interfere with study therapy (e.g. acute leukemias, accelerated/blast-phase chronic myelogenous leukemia, chronic lymphocytic leukemia, Burkitt lymphoma, plasma cell leukemia, or non-secretory myeloma)
* Known primary central nervous system (CNS) malignancy, active or untreated CNS metastases, symptomatic CNS metastases, and/or leptomeningeal disease
* Patients with eczema, psoriasis, lichen simplex chronicus of vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis would be excluded) are permitted provided that they meet the following conditions:

  * Patients with psoriasis must have a baseline ophthalmologic exam to rule out ocular manifestations
  * Rash must cover less than 10% of body surface area (BSA)
  * Disease is well controlled at baseline and only requiring low potency topical steroids (e.g., hydrocortisone 2.5%, hydrocortisone butyrate 0.1%, flucinolone 0.01%, desonide 0.05%, aclometasone dipropionate 0.05%)
  * No acute exacerbations of underlying condition within the last 12 months (not requiring psoralen plus ultraviolet A radiation [PUVA], methotrexate, retinoids, biologic agents, oral calcineurin inhibitors; high potency or oral steroids)
* Any other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications
* Malignancies other than the disease under study within 5 years prior to Cycle 1, Day 1, with the exception of those with a negligible risk of metastasis or death and with expected curative outcome (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer treated surgically with curative intent, or ductal carcinoma in situ treated surgically with curative intent) or undergoing active surveillance per standard-of-care management (e.g. prostate cancer with Gleason score ≤ 6, and prostate-specific antigen [PSA] 10 mg/mL, etc).

Medication-Related Exclusion Criteria:

* Prior treatment with anti-PD-1, and CTLA-4, or anti-a PD-L1 therapeutic antibody or pathway-targeting agents
* Treatment with systemic immunostimulatory agents (including but not limited to interferon [IFN]-a or interleukin [IL]-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to Cycle 1, Day 1
* Concomitant use of another investigational agent and/or treatment with an investigational agent within 4 weeks prior to Cycle 1, Day 1 (or within five half-lives of the investigational product, whichever is longer)
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to Cycle 1, Day 1

  * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled.
  * The use of inhaled corticosteroids or mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed.
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Known hypersensitivity to Chinese hamster ovary cell products or any component of the atezolizumab formulation

Phase I Cohort

* Prior chemotherapy or immunotherapy for metastatic urothelial bladder cancer. Prior neoadjuvant or adjuvant chemotherapy with first progression > 12 months is allowed.
* Any approved anti-cancer therapy within 3 weeks prior to enrollment with the following exceptions:

  * Palliative radiotherapy for bone metastases must be completed > 7 days prior to baseline imaging and > 21 days prior to cycle 1 day 1 of treatment.
  * Hormone replacement therapy or oral contraceptives are permitted
  * Administration of intravesical bacillus Calmette-Guerin (BCG) >4 weeks before Cycle 1, Day 1 is allowed
* Tumor-related pain increased above baseline for 2 weeks and not controlled by a stable dose of opiates
* Uncontrolled pleural effusion, pericardial effusion, or ascites (indwelling drainage catheters allowed)

Phase 2 Cohort

* Prior systemic chemotherapy (prior intravesical therapy is allowed)
* Prior radiation therapy to the bladder
* Any approved anti-cancer therapy within 3 weeks prior to enrollment
* Administration of intravesical bacillus Calmette-Guerin (BCG) >4 weeks before Cycle 1, Day 1 is allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-12-20; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Test the safety of atezolizumab in combination with gemcitabine/cisplatin as assessed by dose limiting toxicity rate. | Participants will be followed for survival until 5 years from treatment completion or until disease recurrence/progression.
  CTCAE version 4.0 will be used for all patients on this trial for evaluation of toxicities during systemic therapy.

SECONDARY OUTCOMES:
Relapse-Free Survival | 3 years
  Relapse-Free Survival by RECIST v1.1 is measured from the time of treatment initiation until the first date that disease progression is objectively documented.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Funt, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (11):
- United States (11):
  - Hartford Healthcare Cancer Institute @ Hartford Hospital, Hartford, Connecticut
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - New York University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Ohio State University, Columbus, Ohio
  - Lehigh Valley Health Network, Allentown, Pennsylvania

REFERENCES:
- [Derived] Funt SA, Lattanzi M, Whiting K, Al-Ahmadie H, Quinlan C, Teo MY, Lee CH, Aggen D, Zimmerman D, McHugh D, Apollo A, Durdin TD, Truong H, Kamradt J, Khalil M, Lash B, Ostrovnaya I, McCoy AS, Hettich G, Regazzi A, Jihad M, Ratna N, Boswell A, Francese K, Yang Y, Folefac E, Herr HW, Donat SM, Pietzak E, Cha EK, Donahue TF, Goh AC, Huang WC, Bajorin DF, Iyer G, Bochner BH, Balar AV, Mortazavi A, Rosenberg JE. Neoadjuvant Atezolizumab With Gemcitabine and Cisplatin in Patients With Muscle-Invasive Bladder Cancer: A Multicenter, Single-Arm, Phase II Trial. J Clin Oncol. 2022 Apr 20;40(12):1312-1322. doi: 10.1200/JCO.21.01485. Epub 2022 Jan 28. PMID 35089812
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm